CLINICAL TRIAL: NCT01589120
Title: Using Videos to Facilitate Advance Care Planning for Patients With Heart Failure
Acronym: VIDEO-HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Colorado, Denver (Other); Vanderbilt University (Other); South Shore Hospital (Other); Brigham and Women's Hospital (Other); Boston Medical Center (Other)
Responsible Party: Principal Investigator, Angelo E. Volandes, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2012-P-000341; 1R01HL107268-01 (NIH)
Record Dates: First submitted 2012-04-28; First posted 2012-05-01 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: CHF
Keywords: CHF; video decision aid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (No Intervention): Verbal description of goals of care reflecting usual care
- Video Arm (Experimental): Video intervention group
  Interventions: Behavioral: Video decision aid

INTERVENTIONS:
Behavioral: Video decision aid — Video decision aid of the goals of care
  Arms: Video Arm

SUMMARY:
The purpose of this study is to compare the decision making of subjects with advanced CHF having a verbal discussion about goals of care compared to subjects using a video.

DETAILED DESCRIPTION:
Aim #1: To compare the impact of the intervention on the distribution of end-of-life knowledge, decisional conflict, and preferences among 248 subjects with advanced heart failure randomly assigned to one of two ACP modalities: 1. a video visually depicting the goals of care along with a patient checklist (intervention, 124 subjects), or 2. usual care, i.e., verbal narrative (control, 124 subjects).

Hypothesis #1: Compared to subjects randomized to the verbal narrative group, subjects randomized to the video intervention will be significantly more likely to:

1a. Have more knowledge about their choices

1b. Have less decisional conflict about their decisions

1c. Opt for comfort care and less likely to choose life-prolonging measures

Aim #2: To compare stability of preferences over time (1, 3, and 6 months), concordance rate of preferences (preferences expressed vs. preferences documented in the medical record - both inpatient and outpatient records), and advance care planning discussions (as reported by the patient), among 248 subjects randomized to the video (N=124) vs. verbal narrative (N=124).

Hypothesis #2: Compared to subjects randomized to the verbal narrative group, subjects randomized to the video intervention will be significantly more likely to:

1a. Have more stable preferences over time

1b. Higher concordance rates

1c. Have had an advance care planning discussion

Aim #3: To compare quality of life, anxiety and depression, referral to hospice, place of death, after death bereavement (caregiver), and resource utilization after 6 months and 1 year (or death) among 248 subjects randomized to the video (N=124) vs. verbal narrative (N=124).

Hypothesis #3: Compared to subjects randomized to the verbal narrative group, subjects randomized to the video intervention will be significantly more likely to:

1a. Have a better quality of life (FACIT-Pal, FACIT-Sp-12)

1b. Have earlier referral to hospice in subjects who die

1d. Die at home or hospice (or inpatient hospice setting) in subjects who die

1e. Have better caregiver bereavement score (for caregiver subjects who die).

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of advanced heart failure as defined by ALL THREE of the following:

   • New York Heart Association Class III or IV (NYHA III or IV) (III: marked limitation in activity due to symptoms, even during less-than-ordinary activity; IV: severe limitations, experiences symptoms while at rest).

   AND
   * Hospitalization for heart failure within the last six months. AND
   * Age greater than or equal to 65.
2. Additionally ONE of the following must be met:

   * According to the attending physician's best judgment the patient's survival is limited to 2 years but may very well be less than 1 year (i.e. the physician would not be surprised if the patient died within one year from any cause) OR
   * Three heart failure hospitalizations in the last year OR
   * One of the following:

     * Two Systolic Blood Pressures < 90 within the last 6 months in the ambulatory setting
     * Na < 130 within the last 6 months
     * NTproBNP > 3,000
     * EGFR < 35
     * High diuretic use (160 mg po Lasix or 100 mg po torsemide or equivalent total daily dose)

Exclusion Criteria:

* New patient
* A transplant or mechanical circulatory support candidate
* Major psychiatric illness as determined by the attending that would make this study inappropriate.
* Any patient that has been excluded for transplant or mechanical circulatory support due to psychological or psychiatric co-morbidities.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2012-04; Primary Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
knowledge | 5 minutes after survey
  knowledge of the goals of care for CHF
preferences | 5 minutes after survey
  preferences for goals of care

SECONDARY OUTCOMES:
decisional conflict | 5 minutes after survey
  decisional conflict regarding decision making
stability | 5 minutes after survey and then at 1, 3, and 6 months
  stability of preferences for goals of care
concordance of preferences | by the end of one year
  concordance of stated preferences with documented preferences in the medical record
advance care planning discussion | by 6 months
  self reported completion of advance care planning discussion
quality of life | after 6 months
  better quality of life using FACIT questionnaire after 6 months
referral to hospice | by one year
  referral to hospice for patients who die
place of death | by one year
  place of death for those patients that die
caregiver bereavement score | by one year
  caregiver bereavement score for those subjects that die

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] El-Jawahri A, Paasche-Orlow MK, Matlock D, Stevenson LW, Lewis EF, Stewart G, Semigran M, Chang Y, Parks K, Walker-Corkery ES, Temel JS, Bohossian H, Ooi H, Mann E, Volandes AE. Randomized, Controlled Trial of an Advance Care Planning Video Decision Support Tool for Patients With Advanced Heart Failure. Circulation. 2016 Jul 5;134(1):52-60. doi: 10.1161/CIRCULATIONAHA.116.021937. PMID 27358437